CLINICAL TRIAL: NCT00713544
Title: A Randomised, Double Blind, Placebo Controlled, Phase IIb Dose Ranging Study (With Open-label Etanercept Treatment Group) to Investigate Efficacy, Safety and Pharmacokinetics of AZD5672 Administered for 12 Weeks to Rheumatoid Arthritis Patients Receiving Methotrexate.
Brief Title: A Proof of Concept and Dose Ranging Study in Patients With Rheumatoid Arthritis
Acronym: ESCAPE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D1710C00009
Record Dates: First submitted 2008-07-09; First posted 2008-07-11 (Estimated); Results first posted 2011-10-03 (Estimated); Last update posted 2011-10-03 (Estimated); Status verified 2011-08

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; RA; AZD5672
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — N-(1-(3-(3,5-difluorophenyl)-3-(4-methanesulfonylphenyl)propyl)piperidin-4-yl)-N-ethyl-2-(4-methanesulfonylphenyl)acetamide; Etanercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1 (Active Comparator)
  Interventions: Drug: Etanercept
- 2 (Experimental): 20mg
  Interventions: Drug: AZD5672
- 3 (Experimental): 50mg
  Interventions: Drug: AZD5672
- 4 (Experimental): 100mg
  Interventions: Drug: AZD5672
- 5 (Experimental): 150mg
  Interventions: Drug: AZD5672
- 6 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD5672 — 20 mg oral, once daily
  Arms: 2
Drug: Etanercept — 50 mg, subcutaneous injection, weekly
  Other Names: Enbrel
  Arms: 1
Drug: Placebo — placebo, oral, once daily
  Arms: 6
Drug: AZD5672 — 50 mg oral, once daily
  Arms: 3
Drug: AZD5672 — 100 mg oral, once daily
  Arms: 4
Drug: AZD5672 — 150 mg oral, once daily
  Arms: 5

SUMMARY:
This study is being carried out to investigate if AZD5672 is effective in treating Rheumatoid Arthritis (RA) and if so how it compares to placebo (a substance which does not have any action) and etanercept (a medicine already available to treat Rheumatoid Arthritis) when added to treatment with methotrexate. The purpose of this study is also to find out which dose of AZD5672 is the most effective at treating RA and to find out how well the body tolerates AZD5672 when taken for up to 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RA with active disease defined as: ≥4 swollen joints and ≥6 tender/painful joints, and either have (blood tests) elevated erythrocyte sedimentation rate (ESR) or C-reactive protein (CRP).
* At least one of the following: documented history of positive rheumatoid factor (blood test), current presence of positive rheumatoid factor (blood test), baseline radiographic erosion, presence of serum anti-cyclic citrullinated peptide antibodies (bloo
* Be receiving either: Oral (tablets) or subcutaneous (injection) methotrexate for at least 6 months prior to randomisation.

Exclusion Criteria:

* Any other inflammatory disease in addition to RA that may interfere with the study (e.g. polymyalgia rheumatica, giant cell arteritis, reactive arthritis, etc).
* Current chronic pain disorders including fibromyalgia and chronic fatigue syndromes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 373 (Actual)
Dates: Start 2008-07; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Layton, Study Director — AstraZeneca; Paul P Tak, MD, PhD, Principal Investigator — University of Amsterdam
Locations (49):
- Bulgaria (3):
  - Research Site, Blagoevgrad
  - Research Site, Plovdiv
  - Research Site, Sofia
- Colombia (3):
  - Research Site, Medellín, Colombia
  - Research Site, Bogotá
  - Research Site, Bucaramanga
- Czechia (7):
  - Research Site, Česká Lípa
  - Research Site, České Budějovice
  - Research Site, Hlučín
  - Research Site, Pardubice
  - Research Site, Prague
  - Research Site, Praha 11 - Chodov
  - Research Site, Zlín
- Hungary (6):
  - Research Site, Békéscsaba
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Kecskemét
  - Research Site, Makó
  - Research Site, Sopron
- Research Site, Siena, SI, Italy
- Research Site, Valmiera, Latvia
- Research Site, Birkirkara, Malta
- Poland (9):
  - Research Site, Bialystok
  - Research Site, Działdowo
  - Research Site, Krakow
  - Research Site, Lublin
  - Research Site, Sopot
  - Research Site, Szczecin
  - Research Site, Torun
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Romania (3):
  - Research Site, Brasov
  - Research Site, Bucharest
  - Research Site, Ploieşti
- Russia (2):
  - Research Site, Saint Petersburg
  - Research Site, Yaroslavl
- Serbia (2):
  - Research Site, Belgrade
  - Research Site, Niška Banja
- Slovakia (3):
  - Research Site, Banská Bystrica
  - Research Site, Bratislava
  - Research Site, Piešťany
- South Africa (3):
  - Research Site, Pretoria, Gauteng
  - Research Site, Durban, KwaZulu-Natal
  - Research Site, Cape Town, Western Cape
- Ukraine (5):
  - Research Site, Donetsk
  - Research Site, Ivano-Frankivsk
  - Research Site, Kiev
  - Research Site, Kyiv
  - Research Site, Simferopol

REFERENCES:
- [Derived] Gerlag DM, Hollis S, Layton M, Vencovsky J, Szekanecz Z, Braddock M, Tak PP; ESCAPE Study Group. Preclinical and clinical investigation of a CCR5 antagonist, AZD5672, in patients with rheumatoid arthritis receiving methotrexate. Arthritis Rheum. 2010 Nov;62(11):3154-60. doi: 10.1002/art.27652. PMID 20662070

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first participant enrolled on 01 July 2008, and the last participant completed the study on 08 April 2009. Participants were recruited from 61 centres in 14 countries in Europe, Southern Africa and South America.
Pre-assignment Details: Male or female adult patients with active rheumatoid arthritis (on background treatment of methotrexate) were randomly assigned to receive AZD5672 at 20, 50, 100 or 150 mg once daily, placebo or etanercept.
  It was planned to randomise approx 360 patients in total, 60 to the open-label etanercept arm and 300 in total to the AZD5672 or placebo arms.
Groups:
- AZD5672 20 mg: AZD5672 20 mg, oral tablets, once daily, double-blinded
- AZD5672 50 mg: AZD5672 50 mg, oral tablets, once daily, double-blinded
- AZD5672 100 mg: AZD5672 100 mg, oral tablets, once daily, double-blinded
- AZD5672 150 mg: AZD5672 150 mg, oral tablets, once daily, double-blinded
- Placebo: Placebo to AZD5672, oral tablets, once daily, double-blinded
- Etanercept: Etanercept 50 mg, subcutaneous injection, once weekly, open-label
Period: Overall Study
Arm/Group | AZD5672 20 mg | AZD5672 50 mg | AZD5672 100 mg | AZD5672 150 mg | Placebo | Etanercept
Started | 52 | 52 | 52 (Participants randomised. One of these participants did not subsequently receive treatment.) | 76 | 65 | 76 (Participants randomised. One of these participants did not subsequently receive treatment.)
Completed | 45 | 46 | 41 | 66 | 57 | 67
Not Completed | 7 | 6 | 11 | 10 | 8 | 9
Not completed — Adverse Event | 5 | 3 | 7 | 7 | 3 | 5
Not completed — Withdrawal by Subject | 2 | 0 | 3 | 2 | 3 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Lack of Efficacy | 0 | 1 | 0 | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0
Not completed — AZ decision - Hepatitis C ab reactive | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Incorrect enrollment | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Hepatotoxicity - not an AE | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD5672 20 mg | AZD5672 50 mg | AZD5672 100 mg | AZD5672 150 mg | Placebo | Etanercept | Total
Number analyzed (Participants) | 52 | 52 | 51 | 76 | 65 | 75 | 371
Age Continuous [Mean (Standard Deviation); unit: Year] | 53 (12.7) | 53 (12) | 54 (10.8) | 53 (10.2) | 53 (10.6) | 54 (9.6) | 53 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 45 | 45 | 67 | 54 | 66 | 322
  Male | 7 | 7 | 6 | 9 | 11 | 9 | 49
Duration of rheumatoid arthritis [Number; unit: participants]
  Duration of rheumatoid arthritis > 5 years | 23 [lower limit 29] | 30 | 25 | 39 | 36 | 48 | 201 [0 to 0]
  Duration of rheumatoid arthritis <= 5years | 29 | 22 | 26 | 37 | 29 | 27 | 170
Disease Activity Score (based on 28 joint counts) (DAS28) [Mean (Standard Deviation); unit: Units on a scale] — Change from baseline in the DAS28 composite score (a measure of RA symptoms including: joint swelling and tenderness; patient's assessment of disease activity; and ESR) after 12 Weeks' treatment. A change of zero indicates no effect of treatment and a negative change of 1.2 indicates a clinically important improvement in symptoms. The DAS scale runs from 0 to 10, with the higher scores indicating worse RA symptoms.
  Units on a scale | 6.6 (0.80) | 6.5 (0.87) | 6.4 (0.72) | 6.3 (0.79) | 6.6 (0.74) | 6.7 (0.80) | 6.5 (0.79)

OUTCOME MEASURES:

1. Primary Outcome: American College of Rheumatology 20 Response (ACR20)
Description: The number of participants with greater to or equal to 20% improvement in the ACR composite score (a measure of RA symptoms including: joint swelling and tenderness; patient's assessment of pain, disease activity and physical function; physician's assessment of disease activity; and CRP) after 12 Weeks' treatment.
Time Frame: 12 weeks
Measure: Number; unit: Participants
Arm/Group | AZD5672 20 mg | AZD5672 50 mg | AZD5672 100 mg | AZD5672 150 mg | Placebo | Etanercept
Number analyzed (Participants) | 52 | 52 | 51 | 76 | 65 | 75
Participants | 20 | 15 | 17 | 34 | 25 | 58

2. Secondary Outcome: American College of Rheumatology 50 Response (ACR50)
Description: The number of participants with greater to or equal to 50% improvement in the ACR composite score (a measure of RA symptoms including: joint swelling and tenderness; patient's assessment of pain, disease activity and physical function; physician's assessment of disease activity; and CRP) after 12 Weeks' treatment.
Time Frame: 12 weeks
Measure: Number; unit: Participants
Arm/Group | AZD5672 20 mg | AZD5672 50 mg | AZD5672 100 mg | AZD5672 150 mg | Placebo | Etanercept
Number analyzed (Participants) | 52 | 52 | 51 | 76 | 65 | 75
Participants | 10 | 5 | 6 | 11 | 6 | 35

3. Secondary Outcome: American College of Rheumatology 70 Response (ACR70)
Description: The number of participants with greater to or equal to 70% improvement in the ACR composite score (a measure of RA symptoms including: joint swelling and tenderness; patient's assessment of pain, disease activity and physical function; physician's assessment of disease activity; and CRP) after 12 Weeks' treatment.
Time Frame: 12 weeks
Measure: Number; unit: Participants
Arm/Group | AZD5672 20 mg | AZD5672 50 mg | AZD5672 100 mg | AZD5672 150 mg | Placebo | Etanercept
Number analyzed (Participants) | 52 | 52 | 51 | 76 | 65 | 75
Participants | 3 | 2 | 3 | 2 | 3 | 12

4. Secondary Outcome: Disease Activity Score (Based on 28 Joint Count) (DAS28)
Description: Change from baseline in the DAS28 composite score (a measure of RA symptoms including: joint swelling and tenderness; patient's assessment of disease activity; and ESR) after 12 Weeks' treatment. A change of zero indicates no effect of treatment and a negative change of 1.2 indicates a clinically important improvement in symptoms. The DAS scale runs from 0 to 10, with the higher scores indicating worse RA symptoms.
Time Frame: Baseline to 12 Weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | AZD5672 20 mg | AZD5672 50 mg | AZD5672 100 mg | AZD5672 150 mg | Placebo | Etanercept
Number analyzed (Participants) | 52 | 52 | 51 | 76 | 65 | 75
Units on a scale | -1.3 (1.27) | -1.1 (1.01) | -1.3 (1.23) | -1.3 (1.15) | -1.1 (1.13) | -2.6 (1.35)

5. Secondary Outcome: Health Assessment Questionnaire - Disability Index (HAQ-DI)
Description: Change from baseline in HAQ-DI (a measure of patients assessment of physical function scored between zero and 3) after 6 months' treatment, calculated as score at 12 Weeks minus score at baseline. A change of zero indicates no effect of treatment and a negative change of 0.22 or greater indicates an improvement in symptoms. The HAQ-DI scale runs from 0 to 3, with higher scores indicating greater disability.
Time Frame: Baseline to 12 Weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | AZD5672 20 mg | AZD5672 50 mg | AZD5672 100 mg | AZD5672 150 mg | Placebo | Etanercept
Number analyzed (Participants) | 52 | 52 | 51 | 76 | 65 | 75
Units on a scale | -0.3 (0.47) | -0.2 (0.48) | -0.2 (0.40) | -0.3 (0.33) | -0.3 (0.47) | -0.5 (0.49)

ADVERSE EVENTS:
Arm/Group | AZD5672 20 mg | AZD5672 50 mg | AZD5672 100 mg | AZD5672 150 mg | Placebo | Etanercept
Serious Adverse Events (participants affected / at risk) | 0/52 | 1/52 | 2/51 | 2/76 | 1/65 | 0/75
Other Adverse Events (participants affected / at risk) | 12/52 | 11/52 | 15/51 | 21/76 | 15/65 | 16/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZD5672 20 mg (N=52) | AZD5672 50 mg (N=52) | AZD5672 100 mg (N=51) | AZD5672 150 mg (N=76) | Placebo (N=65) | Etanercept (N=75)
Hepatitis Cholestatic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Polymyositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZD5672 20 mg (N=52) | AZD5672 50 mg (N=52) | AZD5672 100 mg (N=51) | AZD5672 150 mg (N=76) | Placebo (N=65) | Etanercept (N=75)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 2 | 3 | 2 | 0 | 0
DYSPEPSIA (Gastrointestinal disorders) | 0 | 1 | 3 | 1 | 2 | 0
NASOPHARYNGITIS (Infections and infestations) | 3 | 2 | 4 | 3 | 4 | 4
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 | 1 | 5 | 5 | 1 | 1
BRONCHITIS (Infections and infestations) | 1 | 3 | 1 | 1 | 1 | 5
VIRAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 4 | 0 | 2
ALANINE AMINOTRANSFERASE INCREASED (Infections and infestations) | 4 | 2 | 3 | 3 | 3 | 5
ASPARTATE AMINOTRANSFERASE INCREASED (Infections and infestations) | 2 | 1 | 2 | 3 | 1 | 4
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 3 | 5 | 1
HEADACHE (Nervous system disorders) | 1 | 3 | 2 | 2 | 1 | 1

LIMITATIONS AND CAVEATS:
Hybrid ACR, ACRn, individual ACR components, Erythrocyte sedimentation rate (ESR), Short-form-36 (SF-36), Rheumatoid Arthritis Quality of Life (RAQoL) and Patient Insight Questionnaire (PIQ) did not provide extra information so are not presented

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less